CLINICAL TRIAL: NCT03774134
Title: Five Year Oncological Outcome After Complete Mesocolic Excision for Sigmoid Colon Cancer: a Population-based Cohort Study
Brief Title: Five Year Oncological Outcome After CME for Sigmoid Colon Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Bispebjerg Hospital (Other); Herlev Hospital (Other); Hvidovre University Hospital (Other); Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMELoS2019
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Sigmoid Neoplasms
Keywords: Colon cancer; Surgery; Oncological outcome; Survival
MeSH Terms: conditions — Sigmoid Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CME group: The CME group consisted of patients, who underwent elective CME for sigmoid colon adenocarcinoma at Nordsjaellands Hospital Hillerød from 1 June 2008 to 31 December 2014.
  Interventions: Procedure: Complete mesocolic excision
- Non-CME group: The non-CME group comprised patients having a elective conventional colon cancer resection for sigmoid adenocarcinoma at the other three colorectal centers in the Capital Region of Denmark from 1 June 2008 to 31 December 2013.
  Interventions: Procedure: Conventional colon resection

INTERVENTIONS:
Procedure: Complete mesocolic excision — Based on the principles of CME. The inferior mesenteric artery (IMA) was divided at its origin from the aorta to perform central lymph nodes dissection along the IMA between the aorta and the branching of the left colic artery. Sigmoid resection included the complete sigmoid colon and resection of the upper part of the rectum to ensure sufficient perfusion of the colo-rectal anastomosis. To achieve sufficient distance at the proximal bowel resection margin, parts of the descending colon or even left hemicolectomy were performed at the surgeon's discretion.
  Groups: CME group
Procedure: Conventional colon resection — The patients underwent what was considered standard colon cancer resections in Denmark during the study period.
  Groups: Non-CME group

SUMMARY:
Study based in existing databases investigating the causal oncological treatment effects of complete mesocolic excision on UICC stage I-III sigmoid colon cancer

DETAILED DESCRIPTION:
Population-based cohort study, predominantly prospective based, on the same population as our previously study comparing short-term outcome after CME with conventional colon resections. The COMES database combines the prospectively registered colon cancer database in Hillerød (CME data), and data from the national database of the Danish Colorectal Cancer Group (DCCG) covering patients undergoing conventional resection (non-CME) in the other three centers. The medical records of all the patients in the non-CME group (control group) were reviewed by colorectal surgeons from Hillerød. Data audit for all CME patients was performed by various co-authors employed at the other centers. A similar audit of data for non-CME patients having postoperative complications or recurrence was performed by the co-author representing the department treating the specific patients. Follow-up data were registered prospectively in the medical records of the participating departments during patient follow-up.

Continuous data are presented as median and interquartile ranges, and categorical data as frequencies and proportions. Kruskal-Wallis test and Fisher's exact test were used as appropriate. Death is a competing risk to recurrence and time-to-event analyses were performed as competing risk analyses obtaining the cumulative incidences for recurrence or death using the "cmprsk" R-package.

Unbiased estimation of marginal or population-averaged treatment effects in observational and non-randomized studies can be obtained through different propensity score methods. Inverse Probability of Treatment Weighting (IPTW) uses the propensity score to weight each patient's data based on the inverse probability of receiving the treatment actually received. IPTW gives unbiased estimates of average treatment effects in time-to-event analyses if no differences in observed baseline covariates exist between the treatment groups. To account for baseline differences between patients in the two groups, stabilized weights truncated at the 0.99 interval were calculated using the "IPW" R-package. The following baseline covariates will be used: age, sex, ASA score, neoadjuvant chemotherapy, tumor morphology, perineural invasion, extramural venous invasion, tumor stage, and serosal invasion. All covariates used and UICC stage, two-way interactions, and squared terms of continuous covariates will be assessed for balance between the CME and the non-CME group after IPTW using the "cobalt" R-package. Absolute mean differences in mean (using standardized mean difference) and proportions (using raw mean difference) below 0.1, and variance ratios between 0.5 and 2 will be accepted. Graphical inspection of the distribution of covariates will be also performed.

The cause-specific hazards and overall survival will be analyzed using Cox regression. Binary outcomes were analyzed using logistic regression. Lymph node yield will be analyzed using linear regression after logarithmic transformation. Number of metastatic lymph nodes will be analyzed using negative binominal regression. All analyses of primary and secondary outcomes will be performed after IPTW. The 95% confidence intervals for the estimates from the original Cox regression IPTW analyses will be constructed after 1000 bootstraps with replacement, and a robust sandwich estimator will be used for the logistic regression analyses in order to ensure correct variance estimation.

All available data will be used. Model assumptions will be checked. A p-value below or equal to 0.05 will be considered significant. All analyses will be performed using R statistical software, version 3.5.1 (R Foundation for Statistical Computing, Vienna, Austria).

ELIGIBILITY:
Inclusion Criteria:

* Sigmoid colon cancer was defined as primary adenocarcinomas located in the sigmoid colon (more than 15 cm from the anal verge)
* UICC stage I-III

Exclusion Criteria:

* Synchronous colorectal cancer - even in the sigmoid colon
* No residual tumor in the specimen after neoadjuvant chemotherapy
* Metachronous colorectal cancer
* Resections in Hillerød not performed according to the principles of CME
* Non-macroradical (R2) resections (peroperative assessment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data for all patients undergoing elective surgery for UICC stage I-III colonic adenocarcinoma in the Capital Region of Denmark. The population of this region is approximately 1⋅75 million, more than 30 per cent of the population of Denmark, and it is served by only four public university colorectal cancer centres.
Sampling Method: Non-Probability Sample
Enrollment: 920 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk of recurrence | 5.2 years
  Recurrence diagnosed by CT or positron emission tomography (PET)/CT of thorax and abdomen, chest radiograph and contrast-enhanced ultrasound of the liver, or laparotomy in case of suspicion of recurrence. Histological
  - Page 4 of 6 - verification of radiological findings of metastases during follow-up is not needed if the local multidisciplinary team conference deemed the finding as a recurrence. Metachronous colon tumors diagnosed during follow-up are considered as recurrences only if located in the anastomosis and with the same morphology as the primary tumor.

SECONDARY OUTCOMES:
Overall survival | 5.2 years
  Death by any cause
Short-term mortality | 30 and 90 days
  Death from any cause within 30 and 90 days
Rate of postoperative complications | 60 days
  Patients having surgical and non-surgical postoperative complications and with complications with Clavien-Dindo score of 3b or more
Mesocolic lymph nodes yield | 1 day
  Median number of lymph nodes detected in the specimens and proportion of specimens with 22 or more lymph nodes detected

CONTACTS AND LOCATIONS:
Overall Officials: Claus A Bertelsen, PhD, MD, Study Chair — Department of Surgery, Nordsjaellands Hospital Hillerød

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenberg J, Fischer A, Haglind E; Scandinavian Surgical Outcomes Research Group. Current controversies in colorectal surgery: the way to resolve uncertainty and move forward. Colorectal Dis. 2012 Mar;14(3):266-9. doi: 10.1111/j.1463-1318.2011.02896.x. PMID 22122825
- [Background] West NP, Sutton KM, Ingeholm P, Hagemann-Madsen RH, Hohenberger W, Quirke P. Improving the quality of colon cancer surgery through a surgical education program. Dis Colon Rectum. 2010 Dec;53(12):1594-603. doi: 10.1007/DCR.0b013e3181f433e3. PMID 21178852
- [Background] Hohenberger W, Weber K, Matzel K, Papadopoulos T, Merkel S. Standardized surgery for colonic cancer: complete mesocolic excision and central ligation--technical notes and outcome. Colorectal Dis. 2009 May;11(4):354-64; discussion 364-5. doi: 10.1111/j.1463-1318.2008.01735.x. Epub 2009 Nov 5. PMID 19016817
- [Background] Bokey L, Chapuis PH, Chan C, Stewart P, Rickard MJ, Keshava A, Dent OF. Long-term results following an anatomically based surgical technique for resection of colon cancer: a comparison with results from complete mesocolic excision. Colorectal Dis. 2016 Jul;18(7):676-83. doi: 10.1111/codi.13159. PMID 26476136
- [Background] Bertelsen CA, Neuenschwander AU, Jansen JE, Wilhelmsen M, Kirkegaard-Klitbo A, Tenma JR, Bols B, Ingeholm P, Rasmussen LA, Jepsen LV, Iversen ER, Kristensen B, Gogenur I; Danish Colorectal Cancer Group. Disease-free survival after complete mesocolic excision compared with conventional colon cancer surgery: a retrospective, population-based study. Lancet Oncol. 2015 Feb;16(2):161-8. doi: 10.1016/S1470-2045(14)71168-4. Epub 2014 Dec 31. PMID 25555421
- [Background] Kotake K, Mizuguchi T, Moritani K, Wada O, Ozawa H, Oki I, Sugihara K. Impact of D3 lymph node dissection on survival for patients with T3 and T4 colon cancer. Int J Colorectal Dis. 2014 Jul;29(7):847-52. doi: 10.1007/s00384-014-1885-z. Epub 2014 May 6. PMID 24798631
- [Background] Olofsson F, Buchwald P, Elmstahl S, Syk I. High Tie or not in Resection for Cancer in the Sigmoid Colon? Scand J Surg. 2019 Sep;108(3):227-232. doi: 10.1177/1457496918812198. Epub 2018 Nov 21. PMID 30458672
- [Background] Bertelsen CA, Neuenschwander AU, Jansen JE, Kirkegaard-Klitbo A, Tenma JR, Wilhelmsen M, Rasmussen LA, Jepsen LV, Kristensen B, Gogenur I; Copenhagen Complete Mesocolic Excision Study (COMES); Danish Colorectal Cancer Group (DCCG). Short-term outcomes after complete mesocolic excision compared with 'conventional' colonic cancer surgery. Br J Surg. 2016 Apr;103(5):581-9. doi: 10.1002/bjs.10083. Epub 2016 Jan 18. PMID 26780563
- [Background] Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID 21818162
- [Background] Austin PC, Stuart EA. Moving towards best practice when using inverse probability of treatment weighting (IPTW) using the propensity score to estimate causal treatment effects in observational studies. Stat Med. 2015 Dec 10;34(28):3661-79. doi: 10.1002/sim.6607. Epub 2015 Aug 3. PMID 26238958